CLINICAL TRIAL: NCT00257439
Title: Vitamin Metabolism in Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aalborg University Hospital (Other)
Collaborators: University of Aarhus (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Birn, MD, Aalborg University Hospital
Other Study IDs: VN 2005/44
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Kidney Failure
Keywords: Vitamin B12; Folic Acid
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CKD: Elevated se-creatinine + proteinuria
- Healthy controls: Healthy controls, normal se-creatinine, no proteinuria

SUMMARY:
The purpose of this study is to evaluate the urinary excretion and renal metabolism of vitamins, in particular vitamin B12 and folate, in relation to various renal conditions involving loss of renal function and/or proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the Department of Nephrology, Aalborg Hospital
* Elevated serum creatinine
* Proteinuria
* Informed and written consent

Control subjects:

* Normal serum creatinine and creatinine clearance
* No proteinuria

Exclusion Criteria:

* Vitamin supplementation (exceeding predefined values)
* Renal replacement therapy (dialysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. CKD, proteinuria
  2. Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Birn, MD, PhD, Principal Investigator — Department of Nephrology, Aalborg Hospital
Locations (1):
- Department of Nephrology, Aalborg Hospital, Aalborg, Denmark